CLINICAL TRIAL: NCT01082458
Title: Comparison of Lidocaine and Remifentanil for the Effect on Responses to the Endotracheal Tube During Emergence From General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Jung-Lim Lee / Assistant Professor, Anesthesiology and Pain Medicine
Purpose: Prevention
Other Study IDs: 4-2009-0519
Record Dates: First submitted 2010-03-04; First posted 2010-03-08 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Thyroidectomy
Keywords: Patients scheduled to undergo thyroidectomy
MeSH Terms: interventions — Remifentanil; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: remifentanil / lidocaine — Remifentanil TCI group : target controlled infusion of 2.0ng/ml of remifentanil on end of surgery.
  Lidocaine IV group : Intravenous administration of 1.5mg/kg of lidocaine on end of surgery.

SUMMARY:
Target concentration infusion(TCI) of remifentanil (2.0ng/ml) suppresses the cough induced by endotracheal tube more effectively than intravenous administration of lidocaine (1.5mg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Females older than 20 years old

Exclusion Criteria:

* Patients with acute or chronic respiratory disease, hypertension, gastro-esophageal reflux disease, having preoperative sedatives or mucolytics, and current smoker.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Comparison of lidocaine and remifentanil for the effect on responses to the endotracheal tube during emergence from general anesthesia
  The incidence and the grade of cough during emergence from general anensthesia between remifentanil TCI group and lidocaine IV administration group.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea